CLINICAL TRIAL: NCT04113551
Title: Attention Deficit/Hyperactivity Disorder (ADHD) Medications in Japan: A Retrospective Cohort Study of Label Compliance
Brief Title: A Study of Label Compliance for Attention Deficit/Hyperactivity Disorder (ADHD) Medications in Japan
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108692; PCSESP001604 (Other: Janssen Research and Development, LLC)
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate; Atomoxetine Hydrochloride; Guanfacine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Cohort T1: Methylphenidate (MPH) (Concerta): Analysis of data will be performed for participants who have had first exposure of MPH (Concerta) and who were never exposed to MPH (Ritalin) between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: MPH (Concerta)
- Cohort T2: MPH (Ritalin): Analysis of data will be performed for participants who have had first exposure of MPH (Ritalin) and who were never exposed to MPH (Concerta) between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: MPH (Ritalin)
- Cohort T3: MPH (Concerta and Ritalin): Analysis of data will be performed for participants who have had exposure to Concerta and Ritalin during the time in the cohort between 1 January 2013 and 30 September 2018 and has continuous observation of at least 30 days prior to the exposures.
  Interventions: Drug: MPH (Concerta); Drug: MPH (Ritalin)
- Cohort T4: Atomoxetine (ATO): Analysis of data will be performed for participants who have had first exposure of ATO between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: Atomoxetine (ATO)
- Cohort T5: Guanfacine (GFC): Analysis of data will be performed for participants who have had first exposure of GFC between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: Guanfacine (GFC)
- Cohort T6: MPH (Concerta and Ritalin), ATO, or GFC: Analysis of data will be performed for participants who had have MPH (Concerta or Ritalin), ATO, or GFC first exposure between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure. These are all exposures to any study drug(s) among the participants with an exposure to at least one of the study drugs.
  Interventions: Drug: MPH (Concerta); Drug: MPH (Ritalin); Drug: Atomoxetine (ATO); Drug: Guanfacine (GFC)
- Cohort T7: MPH (Concerta or Ritalin): Analysis of data will be performed for participants who had have MPH (Concerta or Ritalin) first exposure between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior. These are the first exposure to any MPH among the participants with who had some exposure to MPH.
  Interventions: Drug: MPH (Concerta); Drug: MPH (Ritalin)
- Cohort T8: MPH (Concerta) All Exposures: Analysis of data will be performed for participants who have had all exposures of MPH (Concerta) and were never exposed to MPH (Ritalin) between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: MPH (Concerta)
- Cohort T9: MPH (Ritalin) All Exposures: Analysis of data will be performed for participants who have had all exposures of MPH (Ritalin) and were never exposed to MPH (Concerta) between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: MPH (Ritalin)
- Cohort T10: ATO All Exposures: Analysis of data will be performed for participants who have had all exposures of ATO between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: Atomoxetine (ATO)
- Cohort T11: GFC All Exposures: Analysis of data will be performed for participants who have had all exposures of GFC between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure.
  Interventions: Drug: Guanfacine (GFC)
- Cohort T12:MPH(Concerta and Ritalin),ATO,orGFC All Exposures: Analysis of data will be performed for participants who have had all exposures of MPH (Concerta or Ritalin), ATO, or GFC between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure. These are all exposures to any study drug(s) among the participants with an exposure to at least one of the study drugs.
  Interventions: Drug: MPH (Concerta); Drug: MPH (Ritalin); Drug: Atomoxetine (ATO); Drug: Guanfacine (GFC)
- Cohort T13: MPH (Concerta or Ritalin) All Exposures: Analysis of data will be performed for participants who have had all exposures of MPH (Concerta or Ritalin) between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure. These are all exposures to any MPH (Concerta or Ritalin) among the participants with an exposure to MPH (Concerta or Ritalin).
  Interventions: Drug: MPH (Concerta); Drug: MPH (Ritalin)
- Cohort T14: MPH (Concerta and Ritalin) All Exposures: Analysis of data will be performed for participants who have had all exposures of MPH (Concerta and Ritalin) between 1 January 2013 and 30 September 2018 that also has continuous observation of at least 30 days prior to exposure. These are all exposures to any MPH (Concerta or Ritalin) among the participants with an exposure to MPH (Concerta) during the study period and to an exposure to MPH (Ritalin) during the study period.
  Interventions: Drug: MPH (Concerta); Drug: MPH (Ritalin)

INTERVENTIONS:
Drug: MPH (Concerta) — MPH (Concerta) is approved for the indications of ADHD and Narcolepsy in Japan. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from Japan medical data center (JDMC) database.
  Groups: Cohort T12:MPH(Concerta and Ritalin),ATO,orGFC All Exposures; Cohort T13: MPH (Concerta or Ritalin) All Exposures; Cohort T14: MPH (Concerta and Ritalin) All Exposures; Cohort T1: Methylphenidate (MPH) (Concerta); Cohort T3: MPH (Concerta and Ritalin); Cohort T6: MPH (Concerta and Ritalin), ATO, or GFC; Cohort T7: MPH (Concerta or Ritalin); Cohort T8: MPH (Concerta) All Exposures
Drug: MPH (Ritalin) — MPH (Ritalin) is approved for the indication of ADHD in Japan. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from JDMC database.
  Groups: Cohort T12:MPH(Concerta and Ritalin),ATO,orGFC All Exposures; Cohort T13: MPH (Concerta or Ritalin) All Exposures; Cohort T14: MPH (Concerta and Ritalin) All Exposures; Cohort T2: MPH (Ritalin); Cohort T3: MPH (Concerta and Ritalin); Cohort T6: MPH (Concerta and Ritalin), ATO, or GFC; Cohort T7: MPH (Concerta or Ritalin); Cohort T9: MPH (Ritalin) All Exposures
Drug: Atomoxetine (ATO) — Atomoxetine (ATO) is approved for the indication of ADHD in Japan. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from JDMC database.
  Groups: Cohort T10: ATO All Exposures; Cohort T12:MPH(Concerta and Ritalin),ATO,orGFC All Exposures; Cohort T4: Atomoxetine (ATO); Cohort T6: MPH (Concerta and Ritalin), ATO, or GFC
Drug: Guanfacine (GFC) — Guanfacine (GFC) is approved for the indication of ADHD in Japan. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from JDMC database.
  Groups: Cohort T11: GFC All Exposures; Cohort T12:MPH(Concerta and Ritalin),ATO,orGFC All Exposures; Cohort T5: Guanfacine (GFC); Cohort T6: MPH (Concerta and Ritalin), ATO, or GFC

SUMMARY:
The purpose of this study is to document the extent of on-label and off-label use of Methylphenidate (MPH) (Concerta), MPH (Ritalin), Atomoxetine (ATO), and Guanfacine (GFC) in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants have been in the database for greater than or equal to (>=) 30 days
* Have received, between 1 January, 2013 and 30 September, 2018, a prescription for Concerta, Ritalin, Atomoxetine (ATO) or Guanfacine (GFC)

Exclusion Criteria:

- Participants who received an unspecified Methylphenidate (MPH) formulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise of population (participants with attention deficit/hyperactivity disorder [ADHD]) described in the Japan Medical Data Center (JMDC) database which has data available through 1 January 2005 to 30 September 2018.
Sampling Method: Probability Sample
Enrollment: 17418 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Stratified on Age, Sex, and Medication | Up to 5.8 years
  The percentage of participants stratified on age, sex, and medication (Methylphenidate [MPH] [Concerta], MPH [Ritalin], Atomoxetine [ATO], Guanfacine [GFC]) will be reported. The data will be taken from Japan Medical Data Center (JMDC) database for analysis.
Percentage of the Specialty of the Department of the First Prescriber who Prescribe MPH (Concerta), MPH (Ritalin), ATO, or GFC | Up to 5.8 years
  The percentage of specialty of the department of the first prescriber for each first dispensing of each study medication will be reported. The data will be taken from JMDC database for analysis.
Percentage of Participants whose First Prescription for MPH (Concerta), MPH (Ritalin), ATO, or GFC was Associated with an On-label Diagnosis | Up to 5.8 years
  The percentage of participants whose first prescription for MPH (Concerta), MPH (Ritalin), ATO, or GFC was associated with an on-label diagnosis, that is, a diagnosis of Attention Deficit Disorder with Hyperactivity (ADHD) for MPH (Concerta), ATO or GFC; or a diagnosis of narcolepsy for MPH (Ritalin) will be reported. The data will be taken from JMDC database for analysis.
Percentage of Participants who Received More than Maximum Recommended Dose of MPH (Concerta), MPH (Ritalin), Methylphenidate (Concerta and Ritalin), ATO, or GFC | Up to 5.8 years
  The percentage of participants who received more than the maximum recommended dose of MPH (Concerta), MPH (Ritalin), Methylphenidate (Concerta and Ritalin), ATO, or GFC will be reported. The data will be taken from JMDC database for analysis.
Percentage of Participants not Meeting Age Criteria at the Time of Receiving Medication | Up to 5.8 years
  Percentage of participants who at the time of receiving the medication were outside the approved age range will be reported. The data will be taken from JMDC database for analysis.
Percentage of Participants not Meeting Medication Criteria at the Time of Receiving Medication | Up to 5.8 years
  Percentage of participants who at the time of receiving the medication had other contraindications will be reported. The data will be taken from JMDC database for analysis.
Percentage of Participants whose Prescriptions were Consistent with all Aspects of the Label that was Current at the Time of the Prescription | Up to 5.8 years
  Percentage of participants whose prescriptions were consistent with all aspects of the label that was current at the time of the prescription will be reported. The data will be taken from JMDC database for analysis.
Percentage of Participants with Shopping Behavior as a Marker of Misuse of Medications | Up to 5.8 years
  Percentage of participants whose use pattern of MPH (Concerta), MPH (Ritalin), MPH (Concerta and Ritalin) or ATO included prescriptions from three or more departments within any 18-month period will be reported. This describes "shopping behavior", which is a marker for misuse or abuse of medications. The data will be taken from JMDC database for analysis.
Time Trends in Percentage of Participants Compliant with all Label Requirements | Up to 5.8 years
  The time trends in the percentage of participants whose prescriptions complied with all requirements of the label for MPH (Concerta), MPH (Ritalin), MPH (Concerta and Ritalin), ATO, and GFC will be reported. The data will be taken from JMDC database for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (1):
- Janssen Investigative Site, Titusville, New Jersey, United States

REFERENCES:
- [Derived] Fife D, Voss EA, Hardin J, Rofael H, Solomon ID, Ryan PB, Stang P. Medications for attention-deficit/hyperactivity disorder in Japan: A retrospective cohort study of label compliance. Neuropsychopharmacol Rep. 2021 Sep;41(3):385-392. doi: 10.1002/npr2.12191. Epub 2021 Jun 28. PMID 34180161